CLINICAL TRIAL: NCT06481189
Title: A Single-blind Randomized Parallel-group Comparative Study of the Pharmacokinetics, Pharmacodynamics, Safety and Immunogenicity of GNR-086 and Ilaris® After a Single Subcutaneous Administration to Healthy Volunteers at a Dose of 150 mg
Brief Title: A Safety, Pharmacokinetics and Pharmacodynamics Study of GNR-086 and Ilaris® in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AO GENERIUM (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CAN-HVL-I
Record Dates: First submitted 2024-06-20; First posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Healthy Volunteers
Keywords: canakinumab; humanized monoclonal antibodies; safety; pharmacokinetics; equivalence; biosimilar; pharmacodynamics; interleukine-1β
MeSH Terms: interventions — canakinumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GNR-086 (JSC "GENERIUM", Russia) (Experimental): canakinumab biosimilar
  Interventions: Biological: GNR-086
- Ilaris® (Novartis Pharma Stein AG, Switzerland) (Active Comparator): canakinumab
  Interventions: Biological: Ilaris®

INTERVENTIONS:
Biological: GNR-086 — The test drug GNR-086 was administered as a subcutaneous injection at a single dose of 150 mg.
  Other Names: canakinumab
  Arms: GNR-086 (JSC "GENERIUM", Russia)
Biological: Ilaris® — The reference drug Ilaris® was administered as a subcutaneous injection at a single dose of 150 mg.
  Other Names: canakinumab
  Arms: Ilaris® (Novartis Pharma Stein AG, Switzerland)

SUMMARY:
This is a randomized single-blind comparative parallel group study of the safety, pharmacokinetics and pharmacodynamics of GNR-086 and Ilaris® in healthy volunteers. Participants received a single subcutaneous dose of canakinumab 150 mg. The follow up period was 120 days.

DETAILED DESCRIPTION:
GNR-086 (canakinumab) is being developed as a biosimilar to the drug Ilaris®, a lyophilisate for the preparation of solution for subcutaneous administration.

Canakinumab is a recombinant human monoclonal antibody against human interleukine-1β that belongs to the immunoglobulin G1/k (IgG1/k) isotype subclass.

This study is intended for a comparative study of the safety, pharmacokinetics and pharmacodynamics of the drug GNR-086 and the reference drug Ilaris® for the purpose of registration of the drug - GNR-086 (JSC GENERIUM, Russia), 150 mg, lyophilisate for the preparation of solution for subcutaneous administration in the Russian Federation. The study included healthy volunteers aged 18-45 years at the time of signing the informed consent form. The study included a screening period, single administration of study/comparator drug and a follow up period. Allocation of patients to treatment groups was carried out by randomization in a ratio of 1:1 to the study drug and comparator drug. 105 patients (53 to the study drug group and 52 to the comparator drug group) were randomized.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate in the study, obtained from the volunteer before the start of any procedures related to the study;
* Men and women aged 18 to 45 years, inclusive, at the time of signing the informed consent form;
* Verified diagnosis "healthy" (the diagnosis "healthy" is established on the basis of a detailed medical history, in the absence of deviations from normal values during a clinical examination, including measurement of blood pressure, heart rate, respiratory rate, body temperature, as well as laboratory data studies, results of electrocardiography and fluorography);
* Body weight from 50 to 85 kg, body mass index from 18.5 to 28 kg/m2, inclusive.
* Agreement to adhere to adequate methods of contraception during the entire period of participation in the study or for 3 months after administration of the study or reference drug in case of early termination of participation in the study.

Exclusion Criteria:

* Severe chronic diseases, history of seizures;
* Acute infectious diseases less than 4 weeks before administration of the study or reference drug;
* Any history of chronic or recurrent infectious diseases;
* History of tuberculosis;
* Vaccination with any vaccine within 3 months before the administration of the study or reference drug or planned for the period of the volunteer's participation in the study;
* Compounded allergy history; history of hypersensitivity to the active substance or other components of the study or reference drug;
* Pregnancy or breastfeeding period;
* Special lifestyle (work at night, extreme physical activity);
* Deviations of vital signs: systolic pressure less than 100 mm Hg. Art. or more than 130 mm Hg. Art.; diastolic pressure less than 60 mm Hg. Art. or more than 90 mm Hg. Art.; heart rate less than 60 beats/min or more than 90 beats/min;
* Dehydration due to diarrhea, vomiting, or other cause within 24 hours prior to administration of the study or reference drug;
* Taking prescription medications within 28 days or 5 half-lives (whichever is longer) or taking over-the-counter medications/dietary supplements within 14 days prior to study or reference drug administration (occasional use of paracetamol at any time prior to study drug administration is acceptable) or reference drug);
* Blood donation or blood loss (450 ml of blood or more) less than 3 months before the administration of the study or reference drug and/or blood donation in any quantity planned for the period of the volunteer's participation in the study;
* Participation in clinical trials of medicinal products (less than 3 months or 5 half-lives from the study drug, whichever is longer) before administration of the investigational or reference drug of this study;
* Regular alcohol consumption exceeding 5 units. alcohol per week (where each unit is equal to 30 ml of ethyl alcohol or 325 ml of beer), or information about a history of alcoholism, drug addiction, or drug abuse;
* Positive test for the presence of alcohol in exhaled air;
* Smoking more than 5 cigarettes per day for 3 months before this study;
* Positive urine test for the content of narcotic and potent drugs;
* Positive test for hepatitis B, C, HIV or syphilis;
* Any surgical interventions planned during the period of participation in the study;
* Unwillingness or inability to comply with the requirements of this protocol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2023-03-17 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: Area under the plasma concentration versus time curve (AUC) | Day 120
  Analysis of equivalence of area under concentration-time curve from time 0 (predose) extrapolated to infinity (AUC(0-∞) of GNR-086 and Ilaris®
Pharmacokinetics: Peak Plasma Concentration (Cmax) | Day 120
  Analysis of equivalence of Cmax of GNR-086 and Ilaris®

SECONDARY OUTCOMES:
Pharmacodynamics: interleukin-1β (IL-1β) | Day 120
  IL-1β concentration
Pharmacodynamics: Area Under IL-1β Curve (AUC) | Day 120
  Area under the curve "Relative difference in total IL-1β concentration compared to baseline - time"
Proportion of volunteers with adverse events (AE) | Day 120
  The Investigator will carefully monitor each subject throughout the study for any AEs (coded to preferred term and system organ class using the Medical Dictionary for Regulatory Activities [MedDRA])
Immunogenicity | Day 120
  Antidrug antibodies (ADA) level

CONTACTS AND LOCATIONS:
Overall Officials: Oksana A. Markova, MD, Study Chair — JSC GENERIUM
Locations (2):
- Russia (2):
  - State budgetary healthcare institution of the city of Moscow "City Clinic No. 2 of the Moscow Health Department", Moscow
  - Federal State Budgetary Educational Institution of Higher Education "Moscow State Medical and Dental University named after A.I. Evdokimov" of the Ministry of Health of the Russian Federation, Moscow

IPD SHARING:
Plan to Share IPD: No